CLINICAL TRIAL: NCT07276854
Title: Study of a Novel Near-Infrared (NIR) Fluorescent Molecular Probe Based on Humanized Ferritin for the Identification of Benign and Malignant Margins in Gastric Tissue
Brief Title: Novel Humanized Ferritin-based NIR Fluorescent Molecular Probe for Identifying Tumor Margins in Gastric Tissue
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-243
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer; Molecular Imaging
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Indocyanine green-Ferritin (ICG-FTn): Freshly resected gastric cancer specimens were perfused ex vivo via the gastric artery with the targeted probe FTn-ICG solution for about 10 minutes, followed by fluorescence imaging using a DPM system. The results were analyzed to identify tumor regions and delineate tumor margins.
  Interventions: Diagnostic Test: Diagnostic Test: ICG-FTn perfusion solution

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: ICG-FTn perfusion solution — The freshly resected gastric cancer specimens were arterially perfused with ICG-FTn solution and underwent fluorescence imaging.

SUMMARY:
Radical surgery remains the primary treatment for gastric cancer, but intraoperative tumor margin assessment relies on surgeons' visual inspection, limiting accuracy. There is thus an urgent clinical need for real-time visualisation of tumour margins.

In recent years, near-infrared (NIR) fluorescence imaging has emerged as a critical tool for precision tumor resection. However, existing probes like indocyanine green (ICG) lack tumor-targeting specificity. Ferritin (FTn), with its unique nanocage structure, excellent biosafety, and well-defined in vivo behavior, presents an attractive platform for targeted molecular probes.

Yet, translational challenges persist, including animal model limitations and clinical validation bottlenecks. To address this, our study employs freshly resected human gastric tissue in an ex vivo perfusion system, simulating the circulatory dynamics of the humanized ferritin-based probe FTn-ICG in vivo. Using a prospective clinical sample cohort, we aim to validate its diagnostic efficacy in delineating gastric cancer margins, ultimately overcoming the critical barrier of precise tumor boundary identification.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma eligible for radical resection, with histologically verified predominant adenocarcinoma component; Age ≥ 18 years; No gender restriction ; Voluntary participation with written informed consent.

Exclusion Criteria:

* Patients who have received neoadjuvant therapy; Patients deemed ineligible for participation by the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was recruited from the Nanfang Hospital of Southern Medical University in Guangzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The area under the curve (AUC) value of FTn-ICG for diagnostic performance | 2 years
  Pathologists performed histopathological examination of the tumors, while researchers compared the margins identified by pathological results with those predicted by the fluorescence imaging of the probe to calculate the AUC value of ICG-FTn.

SECONDARY OUTCOMES:
Expression of the TfR1 in the tumor | 2 years
  Ability of the imaging system to detect the expression of the TfR1 in tumor tissue.
FTn-ICG distribution in the tumor region | 2 years
  Ability of the imaging system to identify tumor-specific uptake of the targeted probe.
Incidence rates of all adverse events (AEs) | 2 years
  Tissue perfusion adverse events and adverse device events (ADEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No